CLINICAL TRIAL: NCT07299838
Title: Real-World Data for Effectiveness and Safety of Palopegteriparatide in Patients With Chronic Hypoparathyroidism in Greece
Brief Title: Palopegteriparatide in Chronic Hypoparathyroidism
Acronym: PaTHreal
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: G.Gennimatas General Hospital (Other); Alexandra Hospital, Athens, Greece (Other); Theagenio Cancer Hospital (Other Government); 251 Hellenic Air Force & VA General Hospital (Other); Laikο General Hospital, Athens (Other); KAT Hospital of Athens (Unknown); Hellenic Red Cross Hospital (Other); Hippocration General Hospital (Other); Evaggelismos Hospital, Greece (Unknown)
Responsible Party: Principal Investigator, Maria Yavropoulou, Senior Endocrinology Consultant, Laikο General Hospital, Athens
Other Study IDs: 257
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hypoparathyroidism
Keywords: hypoparathyroidism; palopegteriparatide; calcium; phosphate; vitamin D; rhPTH(1-84); real -word-data
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic hypoparathyroidism patients treated with palopegteriparatide: Adult patients with chronic hypoparathyroidism (≥12 months) initiating treatment with palopegteriparatide (TransCon PTH). The cohort includes patients transitioning from conventional therapy (activated vitamin D and calcium supplementation) as well as patients previously treated with rhPTH(1-84). Palopegteriparatide doses were individually titrated based on serum calcium levels and clinical response. Concomitant calcium and activated vitamin D supplementation were adjusted or discontinued according to the treating physician's discretion.

SUMMARY:
This is a multicenter, prospective cohort study conducted across 9 tertiary and university hospitals in the rural area of Athens, which investigates the clinical and biochemical effects of palopegteriparatide (TransCon PTH) in adult patients with chronic hypoparathyroidism (≥12 months). Eligible participants included those transitioning from conventional therapy (activated vitamin D analogs and oral calcium) and those previously treated with rhPTH(1-84). The primary objective was to assess the time to independence from activated vitamin D and calcium supplementation. Secondary objectives included changes in biochemical parameters, incidence of clinically significant hypo- and hypercalcemia during the titration period , and reduction in daily pill burden. Patients received individualized doses of palopegteriparatide with follow-up visits at regular intervals, and safety was monitored throughout the study according to standard clinical practice.

DETAILED DESCRIPTION:
2. Subjects and Methods 2.1 Study Design and Setting

This was a multicenter, prospective cohort study conducted across 9 tertiary and university hospitals in the rural area of Athens. Eligible participants were enrolled from specialized centers experienced in the management of HypoPT between the date that palopegteriparatide was commercially available in Greece (first patient initiating palopegteriparatide was in June 2024) and September 2025. The study included two predefined patient cohorts:

1. Individuals transitioning from conventional therapy (activated vitamin D analogs and calcium supplementation), and
2. Individuals previously treated with rhPTH(1-84) before switching to palopegteriparatide.

2.1.1Participants Adult patients (≥18 years) with a confirmed diagnosis of chronic hypoparathyroidism (HypoPT) of at least 12 months' duration who initiated palopegteriparatide (TransCon PTH)were eligible for inclusion. All participants fulfilled the criteria for PTH replacement therapy as defined by the Hellenic Endocrine Society guidelines.

Diagnosis of chronic HypoPT was established by persistent hypocalcemia in conjunction with inappropriately low or normal serum parathyroid hormone (PTH) concentrations.

Patients were considered eligible for PTH replacement therapy when conventional management failed to achieve optimal biochemical or clinical control, defined by one or more of the following:

* Persistent hypocalcemia or hypocalcemic symptoms despite high-dose oral calcium and active vitamin D supplementation.
* Significant hypercalciuria, nephrolithiasis, nephrocalcinosis, or other renal complications associated with conventional therapy.

To be included in the present analysis, participants were required to have received palopegteriparatide treatment for at least one month prior to data collection or evaluation Exclusion criteria were i) transient postsurgical HypoPT, ii) severe renal impairment (eGFR < 30 mL/min/1.73 m²), iii) active malignancy, iv) Individuals with impaired responsiveness to PTH (pseudohypoparathyroidism)or any disease that might affect calcium metabolism, phosphate metabolism or PTH levels other than hypoparathyroidism, v) other drugs known to influence calcium and bone metabolism (except for activated vitamin D analogs and elemental calcium) such as osteoporosis therapies or glucocorticoids (other than as replacement therapy).

Access to palopegteriparatide in Greece is currently through the National Organization for the Provision of Health Services (EOPYY), which manages reimbursed outpatient and hospital medicines. Medicines for rare diseases or high-cost therapies require pre-approval by relevant health committees. Palopegteriparatide is classified as high-cost medicines and is fully reimbursed upon approval. Continued reimbursement depends on documented treatment response, reductions in conventional therapy burden, control of calcium/urine parameters, and absence of unacceptable adverse events.

2.1.2Treatment Protocol Independent of the last rhPTH(1-84) dose, all patients initiating TransCon PTH were started on 18 µg once daily, as recommended by the manufacturer. The dose was titrated individually based on serum calcium levels, and clinical response, following real-world clinical practice and the product's prescribing information. Concomitant calcium and activated vitamin D supplementation were adjusted or discontinued at the treating physician's discretion to maintain serum calcium within the lower half of the normal range and to minimize hypercalciuria (defined as >250 mg/day in women, >300 mg/day in men, or >4 mg/kg/day in both genders).

2.2 Data Collection and Assessments Baseline data included demographic characteristics, etiology and duration of HypoPT, biochemical parameters (serum calcium, phosphate, magnesium, 25(OH)D, creatinine, and 24-hour urinary calcium), medication use, and comorbidities. Follow-up visits were scheduled at regular intervals according to each center's clinical routine. At each visit, biochemical measurements were recorded, and changes in calcium and vitamin D supplementation, TransCon PTH dose adjustments, and adverse events were documented.

2.3 Ethical Considerations The study protocol was approved by the institutional review boards of all participating centers and conducted in accordance with the principles of the Declaration of Helsinki. Written informed consent was obtained from all participants prior to enrollment.

2.4 Study endpoints 2.4.1 Primary Endpoint The primary endpoint was the time to achievement of independence from activated vitamin D and oral calcium supplementation following initiation of palopegteriparatide. Independence was defined as the absence of any activated vitamin D or calcium supplementation for at least four consecutive weeks, without any increase in the palopegteriparatide dose during that period.

2.4.2 Secondary Endpoints

Secondary endpoints included:

I. The proportion of patients achieving independence from activated vitamin D and calcium within the 14-month observation period.

II. Changes in biochemical parameters (serum calcium, phosphate, magnesium, creatinine, estimated glomerular filtration rate [eGFR], calcium-phosphate product, and 24-hour urinary calcium) between baseline (before initiating palopegteriparatide) and the last follow-up visit.

III. Incidence of clinically significant hypo- and hypercalcemia requiring hospitalization during the study period.

IV. Change in daily pill burden, calculated as the total number of oral calcium and activated vitamin D tablets per day at baseline and last follow-up visit.

2.5. Safety Assessments Safety evaluations were conducted at prespecified intervals, typically every two-three months, in accordance with standard care of clinical practice. Data collected included concomitant medication use, serum biochemistry, hematology, and 25-hydroxyvitamin D levels. Twenty-four-hour urinary calcium excretion was measured periodically. Clinical events such as symptomatic hypo- or hypercalcemia were recorded, and all adverse events deemed treatment-related were documented according to the judgment of the treating physician.

2.6. Statistical Analysis Clinical and biochemical data were analyzed using descriptive and inferential statistics. Categorical variables were presented as absolute numbers and percentages, while continuous variables were expressed as means ± standard deviation (SD) or medians (interquartile range, IQR) where appropriate, depending on data distribution. Normality of distribution was assessed using the Shapiro-Wilk test and inspection of histograms.

To evaluate the effect of palopegteriparatide treatment on biochemical and clinical parameters, within-subject comparisons were performed between baseline (pre-treatment) and the last available follow-up measurement.Τhe paired t-test or the Wilcoxon signed-rank test was applied to compare mean values before and after treatment, as applicable. To explore associations between time to independence from supplements, and biochemical parameters at baseline, duration of the disease or pill burden at baseline, correlation analyses were performed, using Pearson's correlation coefficient (r) or Spearman's rank correlation coefficient (rho), as applicable.

All statistical tests were two-sided, with a significance level of α = 0.05. Confidence intervals (CIs) were two-sided 95%, unless otherwise specified. Analyses were performed using IBM SPSS Statistics (version 28; IBM Corp., Armonk, NY, USA), or equivalent validated statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with a confirmed diagnosis of chronic hypoparathyroidism (HypoPT) of at least 12 months' duration who initiated palopegteriparatide (TransCon PTH)

Exclusion Criteria:

* i) transient postsurgical HypoPT ii) severe renal impairment (eGFR < 30 mL/min/1.73 m²) iii) active malignancy iv) Individuals with impaired responsiveness to PTH (pseudohypoparathyroidism) or any disease that might affect calcium metabolism, phosphate homeostasis, or PTH levels other than hypoparathyroidism v) other drugs known to influence calcium and bone metabolism (except for activated vitamin D analogs and elemental calcium) such as osteoporosis therapies or glucocorticoids other than as replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with a confirmed diagnosis of chronic hypoparathyroidism (HypoPT) of at least 12 months' duration who initiated palopegteriparatide (TransCon PTH)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Time to achievement of independence from activated vitamin D and oral calcium supplementation | From June 2024 (commercial availability of palopegteriparatide in Greece) through September 2025 (end of observation period).
  The primary endpoint was the time to achievement of independence from activated vitamin D and oral calcium supplementation following initiation of palopegteriparatide. Independence was defined as the absence of any activated vitamin D or calcium supplementation for at least four consecutive weeks, without any increase in the palopegteriparatide dose during that period.

SECONDARY OUTCOMES:
Clinical and Biochemical Outcomes Following Palopegteriparatide Treatment in HypoPT Patients | From June 2024 (commercial availability of palopegteriparatide in Greece) through September 2025 (end of observation period).
  I. The proportion of patients achieving independence from activated vitamin D and calcium within the 14-month observation period.
II. To asses changes in albumin corrected calcium levels between baseline and last visit | baseline to last visit within the 14 months of treatmemt
II. To asses changes in phosphate levels between baseline and last visit | baseline to last visit within the 14 months of treatmemt
II. To asses changes in calcium 24 hour urine levels between baseline and last visit | baseline to last visit within the 14 months of treatmemt
II. To asses changes in magnesium levels between baseline and last visit | baseline to last visit within the 14 months of treatmemt

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kassi, M.D, Principal Investigator — Medical School, National and Kapodistrian University of Athens, LAIKO University Hospital of Athens; Symeon Tournis, M.D, Study Director — Laboratory for Research of the Musculoskeletal System "Th. Garofalidis", Medical School, National and Kapodistrian University of Athens, KAT Hospital, 10 Athinas Str, Kifissia, Athens,; Fotini Adamidou, M.D, Study Director — Department of Endocrinology and Diabetes, Hippokratio General Hospital, Thessaloniki, Greece.; Zoe Efstathiadou, MD, Study Director — Department of Endocrinology and Diabetes, Hippokratio General Hospital, Thessaloniki, Greece.; Andromachi Vryonidou, M.D, Study Director — Department of Endocrinology and Diabetes, Hellenic Red Cross Hospital, Athens, Greece.; Polyzois Makras, M.D, Study Director — Department of Endocrinology and Diabetes, Department of Medical Research, 251 Hellenic Air Force General Hospital, Athens, Greece; Dimos Florakis, M.D., Study Director — Department of Endocrinology, Metropolitan General Hospital, Athens, Greece.; Alexandra Chrisoulidou, M.D, Study Director — Department of Endocrinology, Theagenio Cancer Hospital, 54639 Thessaloniki, Greece.; Theodora Stratigou, M.D, Study Director — Department of Endocrinology and First Department of Internal Medicine, 'Evangelismos' General Hospital of Athens, Athens, Greece.; Irene Giagourta, M.D, Study Director — Unit of Endocrinology, and Diabetes Center, 'G. Gennimatas' General Hospital of Athens, Athens, Greece.; Maria Yavropoulou, M.D, Principal Investigator — Medical School, National and Kapodistrian University of Athens, LAIKO University Hospital of Athens
Locations (1):
- Laiko General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Due to participant privacy concerns and institutional policies, individual participant data will not be shared outside the research team

REFERENCES:
- [Result] Khan AA, Guyatt G, Ali DS, Bilezikian JP, Collins MT, Dandurand K, Mannstadt M, Murphy D, M'Hiri I, Rubin MR, Sanders R, Shrayyef M, Siggelkow H, Tabacco G, Tay YD, Van Uum S, Vokes T, Winer KK, Yao L, Rejnmark L. Management of Hypoparathyroidism. J Bone Miner Res. 2022 Dec;37(12):2663-2677. doi: 10.1002/jbmr.4716. Epub 2022 Oct 31. PMID 36161671
- [Result] Khan AA, Bilezikian JP, Brandi ML, Clarke BL, Gittoes NJ, Pasieka JL, Rejnmark L, Shoback DM, Potts JT, Guyatt GH, Mannstadt M. Evaluation and Management of Hypoparathyroidism Summary Statement and Guidelines from the Second International Workshop. J Bone Miner Res. 2022 Dec;37(12):2568-2585. doi: 10.1002/jbmr.4691. Epub 2022 Nov 14. PMID 36054621
- [Result] Rejnmark L, Gosmanova EO, Khan AA, Makita N, Imanishi Y, Takeuchi Y, Sprague S, Shoback DM, Kohlmeier L, Rubin MR, Palermo A, Schwarz P, Gagnon C, Tsourdi E, Zhao C, Makara MA, Ominsky MS, Lai B, Ukena J, Sibley CT, Shu AD. Palopegteriparatide Treatment Improves Renal Function in Adults with Chronic Hypoparathyroidism: 1-Year Results from the Phase 3 PaTHway Trial. Adv Ther. 2024 Jun;41(6):2500-2518. doi: 10.1007/s12325-024-02843-8. Epub 2024 Apr 30. PMID 38691316
- [Result] Siggelkow H, Peschke KA, Tsourdi E, Hofbauer LC, Berr CM, Hahner S, Lottspeich C, Schmidmaier R, Blaschke M. Switch From rhPTH1-84 to TransCon PTH With Individual Dose Adjustment in Adult Hypoparathyroidism-4-Week Results. J Endocr Soc. 2025 Jun 30;9(9):bvaf113. doi: 10.1210/jendso/bvaf113. eCollection 2025 Sep. PMID 40709359
- [Result] Graham T, Shoback DM, Abbott L, Lubitz S, Edelson G, Haider A, Ing SW, Rothman MS, Cusano NE, Zhao C, Ukena J, Schneider M, Sibley CT, Rubin MR. Early U.S. Real-World Treatment Patterns and Outcomes in Palopegteriparatide Treatment for Patients With Hypoparathyroidism. Endocr Pract. 2025 Dec;31(12):1568-1575. doi: 10.1016/j.eprac.2025.08.008. Epub 2025 Aug 20. PMID 40846304
- [Result] Karpf DB, Pihl S, Mourya S, Mortensen E, Kovoor E, Markova D, Leff JA. A Randomized Double-Blind Placebo-Controlled First-In-Human Phase 1 Trial of TransCon PTH in Healthy Adults. J Bone Miner Res. 2020 Aug;35(8):1430-1440. doi: 10.1002/jbmr.4016. Epub 2020 Apr 16. PMID 32212275
- [Result] Khan AA, Rubin MR, Schwarz P, Vokes T, Shoback DM, Gagnon C, Palermo A, Marcocci C, Clarke BL, Abbott LG, Hofbauer LC, Kohlmeier L, Pihl S, An X, Eng WF, Smith AR, Ukena J, Sibley CT, Shu AD, Rejnmark L. Efficacy and Safety of Parathyroid Hormone Replacement With TransCon PTH in Hypoparathyroidism: 26-Week Results From the Phase 3 PaTHway Trial. J Bone Miner Res. 2023 Jan;38(1):14-25. doi: 10.1002/jbmr.4726. Epub 2022 Nov 12. PMID 36271471
- [Result] Khan S, Khan AA. Chronic Hypoparathyroidism-Current and Emerging Therapies. Endocr Pract. 2025 Nov;31(11):1478-1487. doi: 10.1016/j.eprac.2025.07.011. Epub 2025 Jul 16. PMID 40680836
- [Result] Pasieka JL, Wentworth K, Yeo CT, Cremers S, Dempster D, Fukumoto S, Goswami R, Houillier P, Levine MA, Pasternak JD, Perrier ND, Sitges-Serra A, Shoback DM. Etiology and Pathophysiology of Hypoparathyroidism: A Narrative Review. J Bone Miner Res. 2022 Dec;37(12):2586-2601. doi: 10.1002/jbmr.4714. Epub 2022 Nov 23. PMID 36153665
- [Result] Kassi E, Adamidou F, Yavropoulou MP, Anastasilakis AD, Makras P, Vryonidou A, Tournis S. Diagnosis and management of hypoparathyroidism: recommendations of the working group of the Bone Section of the Hellenic Endocrine Society. Hormones (Athens). 2025 Dec;24(4):913-922. doi: 10.1007/s42000-025-00693-9. Epub 2025 Jun 27. PMID 40576884
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40576884/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36153665/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40680836/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36271471/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32212275/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40846304/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40709359/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38691316/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36054621/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36161671/